CLINICAL TRIAL: NCT04281277
Title: Relation Between Mean Arterial Pressure and Renal Resistive Index in the Early Phase of Septic Shock
Acronym: SEPSIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49RC19_0236
Record Dates: First submitted 2020-02-17; First posted 2020-02-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2022-10

CONDITIONS: Septic Shock
Keywords: renal resistive index; mean arterial pressure
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low target group (Active Comparator): target of mean arterial pressure(MAP) at 65-70 mmHg.
  The therapeutic means used to obtain the MAP objectives within each group (increase in catecholamines and / or volume expansion) are left to the discretion of the clinician, in accordance with the recommendations.
  Interventions: Device: increase of mean arterial pressure at 65-70 mmHg.
- high target group (Experimental): target of mean arterial pressure (MAP) at 80-85 mmHg.
  The therapeutic means used to obtain the MAP objectives within each group (increase in catecholamines and / or volume expansion) are left to the discretion of the clinician, in accordance with the recommendations.
  Interventions: Device: increase of mean arterial pressure at 80-85 mmHg.

INTERVENTIONS:
Device: increase of mean arterial pressure at 80-85 mmHg. — increase of mean arterial pressure at 80-85 mmHg (with catecholamines or volemic expansion).
  Arms: high target group
Device: increase of mean arterial pressure at 65-70 mmHg. — increase of mean arterial pressure at 65-70 mmHg (with catecholamines or volemic expansion).
  Arms: low target group

SUMMARY:
This study evaluates if improvement of renal resistive index when mean arterial pressure increase (at 65 mmHg to 85 mmHg) in early phase of septic shock is predictive of better renal survival.

DETAILED DESCRIPTION:
Learned societes (survival sepsis campaign and ESICM) are currently recommending a mean arterial pressure (MAP) target at 65 mmHg in septic shoc with a potential increase to 85 mmHg in patients with medical history of arterial hypertension.

A high renal resistive index on the first day of septic shock was associated with acute renal failure more frequently on the 5th day. A decrease in the renal resistance index was also objectified during the increase in MAP.

The main objective of this trial is to study the relationship between the improvement of the resistance index during a test of increase in average blood pressure during septic shock and the improvement of renal function

In this interventional monocenter trial, we will measure the renal resistive index after stabilization of the MAP at 65 mmHg for two hours, then after 2 hours of stabilization at 85 mmHg. This part allows us to define the patients "responding" to the renal resistive index (improvement of the resitive renal index when the MAP increases).

Then, patients will be randomized into two groups :

* first group with a MAP target at 65 mmHg
* second group with a MAP target at 85 mmHg. There will be a stratification on the responder character to the renal resistance index.

Finally, we will assess renal function on the 7th day (with the assessment of serum creatinine and the change of stage of the KDIGO classification)

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 ans)
* Admitted to the intensive care unit of Angers with
* arterial hypotension requiring the etablishment of catecholamines
* In a context of proven or suspected sepsis, whaterver the cause of this infection.
* norepinephrine dose ⩾ 0.1µg/kg/min
* After 2 hours of stabilization at 65 mmHg of mean arterial pressure

Exclusion Criteria:

* Pre-existing chronic renal failure (glomerular filtration rate < 60 mL/min with MDRD)
* Solitary kidney (anatomical or functional)
* History of united or bilateral stenosis of the renal arteries
* decision to stop or limit treatment
* patient with an emergency indication of renal replacement therapy (severe hyperkalemia, severe metabolical acidosis with pH <7.15, acute pulmonary edema due to fluid overload resulting in severe hypoxemia, serum urea concentration > 40 mmol/l and oliguria/anuria > 72 h.)
* pregnant, lactating or parturient woman
* patient deprived of liberty by judicial or administrative decision
* patient with psychiatric compulsory care
* patient subject to legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
changes of KDIGO stage | Inclusion and day 7
  modification of the KDIGO classification stage (estimated based on serum creatinine and diuresis) between the group with low target of mean arterial pressure ( 65-70 mmHg) and high target MAP (80-85 mmHg)

SECONDARY OUTCOMES:
Renal resistive index | Inclusion, and 2 hours of mean arterial pressure stabilized at 85 mmHg and every day (day 1 to day 7)
  We will assess the evolution of the renal resistive index during an increase in the target of MAP in the early phase of septic shock . We will assess the evolution of renal resistive index according to the comorbidities, as a function of time in septic shock, according to the hemodynamic data, according to quantity of filling solution administered and catecholamine doses
Collection of all adverse event | Day 1 to day 7
  Difference in sides effects between target at 65-70 mmHg of MAP and 80-85 mmHg.
amount of fluids (unit = L or L/day) | Inclusion, day 1 to day 7
catecholamines free days | day 1 to day 7
extra renal replacement free days | Daily to day 1 to day 7, at day 28 and day 90
  Difference in need of renal replacement therapy between the group of 80-85mmHg and the groupe 65-70 mmHg, depending on the responder character
Number of day with supportive care in intensive care unit (renal replacement therapy, mechanical ventilation, extracorporeal membrane oxygenation) | Collection daily between Day 1 and Day 7, at Day 28.
  Quantification of the number of days with supportive care (catecholamine,renal replacement therapy, mechanical ventilation, extracorporeal membrane oxygenation)
Number of day in intensive care unit | Collection at Day 28 and Day 90
  Quantification of the number of days hospitalized in intensive care unit
Number of day in hospital | Collection at Day 28 and Day 90
  Quantification of the number of days hospitalized.
hemodynamic data collected by swan ganz or PICCO catheter | Inclusion and at 2 hours, daily between Day 1 and Day 7
quantity of nephrotoxic drugs | Inclusion and daily between Day 1 and Day 7.
serum creatinine (unit = µmol/L) | Inclusion and daily between Day 1 and Day 7
Diuresis (unit = mL per day) | Daily between day 1 and day 7
Survival at day 28 | patient status (live or dead) at day 28
Survival at day 90 | patient status (live or dead) at day 90
Skin recoloration time evolution | Inclusion and at 2 hours, daily between Day 1 and Day 7
  measurement onto the right index finger by a standardized method after 2 hours of stabilization at 65 mmHg and after 2 hours of stabilization at 85 mmHg.
Skin recoloration time evolution | Inclusion and at 2 hours, daily between Day 1 and Day 7
  measurement onto the right index fingerby a standardized method depending on the randomization group.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ASFAR, MD PHD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers. Médecine Intensive Réanimation et médecine hyperbare, Angers, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).